CLINICAL TRIAL: NCT03618680
Title: Fatigue and Sleep in Children and Adolescents With Juvenile Idiopathic Arthritis: A Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ela Tarakci, Principal Investigator, Assoc.Dr., Istanbul University
Other Study IDs: A29/03.Feb.2015
Record Dates: First submitted 2018-07-24; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Fatigue; Juvenile Idiopathic Arthritis
Keywords: Sleep
MeSH Terms: conditions — Fatigue; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aims of this study is to primarily investigate fatigue and sleep and to secondarily examine possible relationships between disease activity, pain and functional ability in Turkish children and adolescents with Juvenile Idiopathic Arthritis (JIA).

DETAILED DESCRIPTION:
Children with JIA become fatigued easily, experience joint inflammation, pain, limited mobility and report poor sleep quality and daytime sleepiness . It is reported in the literature that children with JIA suffer from poor sleep, parasomnias, daytime sleepiness, sleep fragmentation, cyclic alternating patterns increase, and sleep-disordered breathing compared to healthy children. Sleep was disturbed in almost half of the patients with both JIA and juvenile dermatomyositis, and that sleep disturbance and fatigue were both correlated with disease activity. Increased pain is associated with more sleep disturbance and more fatigue, and these appear to negatively influence quality of life.

So, in this study, fatigue and sleep in Turkish patients with JIA will be investigated by using specific surveys and also secondarily it will be examined possible relationships between disease activity, pain and functional ability in children and adolescents with JIA.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria consisted of a diagnosis of JIA according to the International League of Associations for Rheumatology (ILAR) criteria (13), being aged between 6 - 18 years, and being able to read and write in the Turkish language. All patients were diagnosed as JIA 6 months prior to the study.

Exclusion Criteria:

* Patients were excluded from study if they had a second rheumatic or another chronic disease, a history of mental deficit or psychological problem or no acceptance for participation in the study by their families.

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients attending the outpatient clinic of the Department of Pediatric Rheumatology, Medical Faculty of Cerrahpasa, Istanbul University, were recruited between February 2015 and December 2015 to participate in this study. All participants signed informed consent forms. The participants were volunteers who were examined by the pediatric rheumatologist who participated in the present study.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory-Multidimensional Fatigue Scale | baseline
  Pediatric Quality of Life Inventory-Multidimensional Fatigue Scale" (PedsQL-F) is a valid and reliable tool, and can be used to measure symptom-specific fatigue among patients with JIA . Fatigue symptoms will be assessed by the PedsQL-F which is an 18-item questionnaire and is designed to measure child and parent's perception of fatigue in pediatric patients and comprises the general fatigue scale (6 items), sleep/rest fatigue scale (6 items) and cognitive fatigue scale (6 items). Higher scores indicate higher quality of life.
Pittsburgh Sleep Quality Index | baseline
  Sleep quality will be evaluated with Pittsburgh Sleep Quality Index (PSQI). PSQI is a 23 item questionnaire that generates scales reflecting daytime dysfunction, sleep latency, disturbance, duration, quality and efficiency. As the score increases, sleep quality decreases and daytime dysfunction due to sleep quality disorder increases. PSQI is composed of three main scores: total PSQI score, PSQI sub-scores and sleep quality status score. Each component is scored from 0 to 3, leading to a global PSQI score between 0 and 21, with higher scores indicating lower quality of sleep.

SECONDARY OUTCOMES:
Childhood Health Assessment Questionnaire | baseline
  Functional ability will be assessed using The Turkish version of the Childhood Health Assessment Questionnaire (CHAQ). CIn 8 activities (dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities), a number of questions were answered and scored on a scale of 0 - 3, where 0 = able to do with no difficulty, 1 = able to do with some difficulty, 2 = able to do with much difficulty, and 3 = unable to do. The mean of the 8 scores identified the CHAQ score (range, 0 - 3).